CLINICAL TRIAL: NCT04138316
Title: CandeSpartan Study Candesartan Spanish Response-prediction and Tolerability Study Observational Study on Response Predictors and Tolerability of Candesartan in Usual Clinical Practice
Brief Title: CandeSpartan Study. Candesartan Spanish Response-prediction and Tolerability Study
Acronym: CandeSpartan
Status: Completed | Type: Observational
Sponsor: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Principal Investigator, David García Azorín, Principal investigator, Hospital Clínico Universitario de Valladolid
Other Study IDs: PI 19-1452
Record Dates: First submitted 2019-10-07; First posted 2019-10-24 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Migraine; Head Pain
Keywords: headache disorders
MeSH Terms: conditions — Migraine Disorders; Headache; Headache Disorders | interventions — candesartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Migraine patients
  Interventions: Drug: Candesartan

INTERVENTIONS:
Drug: Candesartan — Treatment with Candesartan

SUMMARY:
Observational, prospective, descriptive, open study on response predictors and tolerability of Candesartan in patients >18 years with episodic or chronic migraine with prior failure of three or more preventive drugs. Patients will receive Candesartan the same manner and intensity if they were not enrolled in the study. Vital signs, clinical variables and adverse events will be monitored.

Primary endpoint will be to determine demographic and clinical factors associated with a 50% reduction in the frequency of headache days per month between weeks 20 and 24 compared with baseline.

DETAILED DESCRIPTION:
CandeSpartan Study Candesartan Spanish Response-prediction and Tolerability study

Observational study on response predictors and tolerability of Candesartan in usual clinical practice

INTRODUCTION:

Migraine is a neurological disease with a prevalence of 14% of the population 1, 2. It is the second most disabling disease in terms of years of life lived with disability, especially in the age group between 15 and 49 years3. Migraine is also the headache the most frequently seen in neurology consultations and headache units4.

Since the 1970s, numerous preventive drugs have been developed. One of the problems is that many of these drugs come from other indications, such as depression, epilepsy or hypertension5. Nowadays, clinical practice guidelines base the indication mainly on the level of evidence6, which, given the age and scarcity of these studies, is limited. Although the new drugs are based on clinical trials according to the current methodology, they are unlikely to be indicated in patients who have not tried any preventive treatment.

Candesartan is an angiotensin-2 receptor antagonist drug that has shown efficacy in episodic migraine mainly in two clinical trials compared to placebo, using a 16 mg daily dose. The first study showed a monthly headache days reduction of 4.9 days of (standard deviation 10.6) in episodic migraine patients that had previously failed to none or one preventive, with 2-6 episodes of headache per month at baseline7. The second study had three arms, including propranolol and placebo showing a montly headache days reduction of -2.91 days (standard deviation 1.06) and showing no-inferiority with respect to propranolol8.

Spanish official headache guidelines recommend Candesartan use in patients with migraine with and without aura, particularly if they have hypertension or comorbid depression6. In some international prestige centers, it is the first choice drug. In habitual clinical practice, one aspect that limits its use is tolerability, being frequent the presence of hypotension and dizziness, even at the dose of 8mg, frequently used in our environment9. In the studies carried out, there were adverse effects in 45-50% of the patients and in 10% of patients was a reason for treatment discontinuation 7, 8.

The aim of our study is to evaluate which clinical factors are associated with a better therapeutic response or a worse tolerability in usual clinical practice.

Hypothesis The therapeutic response and tolerability to candesartan may be influenced by individual factors or related to the evolution of migraine.

PATIENTS AND METHODS:

Design:

Multicentric, prospective, observational, descriptive, open, study of the response and tolerability predictors of candesartan in migraine patients.

Eligibility:

Inclusion criteria:

Diagnosis of migraine (episodic or chronic) according to the International Classification of headache Disorders (ICHD), 3rd version, criteria10.

Being treated with Candesartan under the criteria of the physician and according to local guidelines.

Age >18 years. More than 4 days of headache per month in the preceding 3 months. More than 1 year of migraine evolution. Beginning of migraine before the age of 50. Ability to provide informed consent.

Exclusion criteria:

Previous failure of three or more preventive drugs in accordance with the definition provided below.

Concomitant use of another preventive drug or use of it in less than 5-half lives of the drug.

History of another active primary headache with a periodicity considered frequent according to the International Classification of Headache disorders, that is, more than 10 days per month at the time of screening or the basal period.

Continuous or daily headache in the month prior to inclusion in the study. Pregnancy or breastfeeding. Any relevant cardiovascular conditions. Kidney diseases. Hyperkaliemia. Use of another concomitant preventive. Previous use of candesartan. Current use of another Angiotensin Conversing Enzime Inhibitor or Angiotensin-II receptor antagonist.

Alcoholism or drug use.

Concomitant treatment:

The study will not interfere in the current practice, participants will receive the candesartan in the same manner and intensity if they were not enrolled in the study.

Patients will be allowed to use their usual symptomatic treatment as usual. The number of days of symptomatic treatment and the number of use of triptans will be reflected.

The concomitant drugs with potential use as a preventive according to National Clinical Practice guidelines (gabapentin, pregabalin, tricyclic antidepressants, duloxetine, valproic acid, phenytoin, lamotrigine, topiramate, botulinum toxin, anti-CGRP antibodies, beta-blockers, lisinopril) will not be permitted.

Treatment failure shall be defined as insufficient efficacy at a sufficient dose and for an adequate duration or withdrawal due to adverse effects of a drug present in the national headache guidelines.

Intervention and visits:

The visits will be carried out in the Headache Units of the participating centers. At the baseline visit, investigators will review that patients meet all inclusion criteria and none exclusion criteria. In accordance with the Good Clinical Practice guidelines12, a clear explanation will be given of the objective of the study, the role of the participant and the complete absence of risks that the study pose, due to the observational nature. The participant will be provided with a contact telephone number where he or she can contact in the event of an incident that want to refer to the investigators. The informed consent will be signed and a copy given to the participant.

During the initial visit, the monthly headache days at baseline will be gathered, including the number of days of intense pain, the number of days of taking symptomatic medication, the number of days of taking triptans and the number of visits to the emergency department. A number of demographic and clinical variables (described below) will be reviewed. The patient will be asked to make a prospective record of his or her days of headache as well as the intensity of headache and the use of medication in a standardized diary (appendix) for thirty-six weeks. The presence of possible adverse effects will be detailed. The patient will be evaluated and both basal blood pressure and heart rate will be measured. Headache Impact Test (HIT-6) and Hospital Anxiety and Depression Scale (HADS), Allodynia Symptom Checklist (ASC-12) scales will be administered.

Administration of candesartan:

Participants will receive candesartan in the same manner and intensity as if they would not be enrolled in the study, according to the Spanish national guidelines.

A follow up visit will be done at week 12 to analyze response to candesartan and the possibility of adverse effects. Physicians will modify candesartan dose according to their criteria and the local guidelines. Treatment response will be analyzed during the third visit, at week 24.

Study variables:

Demographic variables:

Sex, current age, age of onset, type of migraine (episodic/chronic), months of evolution of chronic migraine, weight, height, overweight (determined according to the CUN-BAE scale).

Clinical variables:

Presence of aura, bilateral or unilateral predominance, headache intensity (0-10 verbal analogue scale), presence of allodynia (ASC-12 scale), prior history of psychiatric comorbidity (anxiety, depression), impact of headache (HIT-6 scale score).

Headache days per month, intense headache days per month, emergency department visits per month, medication days per month, triptan days per month.

Previous preventive drugs: drug, maximum dose, time of use, presence of adverse effects, response rate (0-30, 30-50, 50-75 or 75-100%).

Blood pressure (mmHg), heart rate (beats per minute).

Safety variables:

Dizziness, tiredness, reduced physical capacity, nausea, constipation, sleep disturbance, sexual dysfunction and paresthesias.

Monitoring of adverse effects:

The patient will spontaneously report the presence of an adverse effect and will also be asked through a structured questionnaire during each visit (appendix). The severity of the adverse effect and the relationship with the study drug with the drug will be detailed and described by the investigator.

Follow-up:

Each patient will use a prospective monthly calendar that will facilitate a correct recording of the characteristics of the headache, including frequency, intensity, need of symptomatic drugs and presence of any adverse events.

During each visit, presence of adverse effects such as pain, sensation of contracture or discomfort will be systematically evaluated. Spontaneous reporting of adverse effects will be allowed and also direct questions will be asked.

OBJECTIVES:

Main objective11:

To determine which demographic or clinical variables present at baseline are associated with a 50% reduction in the frequency of headache days per month between weeks 20 to 24 compared with baseline in a regression analysis.

Secondary objectives:

To determine which demographic and clinical variables present at baseline are associated with a greater reduction in the frequency of headache days per month between weeks 20 to 24 compared with baseline in a regression analysis.

To determine frequency and type of adverse effects related with candesartan through study completion, an average of 24 weeks.

To evaluate percentage of patients that discontinues candesartan due to adverse events through study completion, an average of 24 weeks.

To evaluate percentage of patients that present a 50% response rate to candesartan in headache day reduction evaluated in the period between weeks 20 to 24 compared with baseline.

To evaluate percentage of patients that present a 50% response rate to candesartan in headache day reduction evaluated in the period between weeks 8 to 12 compared with baseline.

To evaluate percentage of patients that present a 30% response rate to candesartan in headache day reduction evaluated in the period between weeks 20 to 24 compared with baseline.

To evaluate percentage of patients that present a 30% response rate to candesartan in headache day reduction evaluated in the period between weeks 8 to 12 compared with baseline.

To evaluate percentage of patients that present a 75% response rate to candesartan in headache day reduction evaluated in the period between weeks 20 to 24 compared with baseline.

To evaluate percentage of patients that present a 75% response rate to candesartan in headache day reduction evaluated in the period between weeks 8 to 12 compared with baseline.

To evaluate percentage of patients that present a 100% response rate to candesartan in headache day reduction evaluated in the period between weeks 20 to 24 compared with baseline.

To evaluate percentage of patients that present a 100% response rate to candesartan in headache day reduction evaluated in the period between weeks 8 to 12 compared with baseline.

To evaluate headache days reduction in the period between weeks 20 to 24 compared with baseline.

To evaluate headache days reduction in the period between weeks 8 to 12 compared with baseline.

To evaluate intense headache days reduction in the period between weeks 20 to 24 compared with baseline.

To evaluate intense headache days reduction in the period between weeks 8 to 12 compared with baseline.

To evaluate acute medication days reduction in the period between weeks 20 to 24 compared with baseline.

To evaluate acute medication days reduction in the period between weeks 8 to 12 compared with baseline.

To evaluate change in HIT-6 scale in the period between weeks 20 to 24 compared with baseline.

To evaluate change in HIT-6 scale in the period between weeks 8 to 12 compared with baseline.

To evaluate change in HADS scale in the period between weeks 20 to 24 compared with baseline.

To evaluate change in HADS scale in the period between weeks 8 to 12 compared with baseline.

To evaluate change in heart rate (in beats per minute) in the period between weeks 20 to 24 compared with baseline.

To evaluate change in heart rate (in beats per minute) in the period between weeks 8 to 12 compared with baseline.

To evaluate change in systolic blood pressure (in mmHg) in the period between weeks 20 to 24 compared with baseline.

To evaluate change in systolic blood pressure (in mmHg) in the period between weeks 8 to 12 compared with baseline.

To evaluate change in diastolic blood pressure (in mmHg) in the period between weeks 20 to 24 compared with baseline.

To evaluate change in diastolic blood pressure (in mmHg) in the period between weeks 8 to 12 compared with baseline.

STUDY DESIGN

Sample size:

For calculation of sample size we used the combined data from both studies, in which, through analysis by intention to treat, the 50% response rate in the group treated with candesartan was 18/57 and 24/66, for a combined response rate of 42/123=34.1%. In the placebo group the 50% response rate in the placebo group was 1/57 and 14/64, for a combined ratio of 15/121=12.4%.

Randomization:

This is an open, not controlled with placebo study.

Stratification:

There will be no stratification of patients. Regression analysis will be performed to evaluate factors associated with better response or worse tolerability.

Statistical aspects:

An anonymous database will be created in which the identity of the patient will be dissociated from the rest of the data. SPSS statistics package will be used for statistical analysis. Analyses will be performed both by intention to treat and per protocol, the primary objective being determined by intention to treat.

The main variable will be calculated by evaluating percentage of patients in whom the number of headache days per month, evaluated between weeks 20-24, is at least 50% lower than the number of headache days per month in the baseline period, before the use of candesartan.

Logistic regression analysis and linear regression will be performed depending on the type of variable and those associated variables with a value of p<0.05 will be selected. In addition, a multivariate regression analysis will be carried out in which all variables with a p<0.015 will be included and a second analysis will be carried out in which the number of days of reduction with respect to the baseline situation between weeks 20 and 24 will be used as a variant.

Factors associated with the presence of adverse effects will be analyzed by logistic or linear regression analysis. 30%, 75% and 100% response rate analysis will also be performed.

To evaluate the reduction in days of pain, the mean number of days of pain between weeks 20-24 and the baseline period will be compared. It will be evaluated if the distribution is normal using the Kolmogorov-Smirnov test and if appropriate, the Student t test will be performed for paired samples; using the Mann-Whitney U test in case the distribution is not normal. The analysis will be repeated for the period between weeks 8-12 and weeks 32-36. The same analysis will also be done to determine the change in the average number of days of severe pain and days of use of symptomatic medication. The mean score on the HIT-6 and HADS scales over the same periods and the change in heart rate and blood pressure will also be compared. The Bonferroni method will be used to correct for multiple comparisons. In the comparison of qualitative variables, the Chi-square test or the exact Fisher test in non-parametric variables will be used. An intermediate analysis will be carried out when 50% of the patients have been recruited.

The management of lost data will be done by imputation in a worse-case scenario. Missing days will be considered days with pain and treatment.

Ethical and legal aspects:

Eligible patients will be exposed to the possibility of participating in the study and if they accept, they will be explained in detail the objective, the procedure and what their participation consists of. If they accept, they must sign an informed consent12. In the event of refusing participation or revoking consent, patients may continue their usual treatment and care process without any modification or conditions. They will be free to refuse to participate in the study or to suspend their collaboration whenever they wish, with no impact on their future medical care.

An anonymized database will be created and stored in the hospital of the principal investigator with the list of participants and personal data dissociated and separated from it.

ELIGIBILITY:
Inclusion criteria:

Diagnosis of migraine (episodic or chronic) according to the International Classification of headache Disorders (ICHD), 3rd version, criteria10.

Being treated with Candesartan under the criteria of the physician and according to local guidelines.

Age >18 years. More than 4 days of headache per month in the preceding 3 months. More than 1 year of migraine evolution. Beginning of migraine before the age of 50. Ability to provide informed consent.

Exclusion criteria:

Previous failure of three or more preventive drugs in accordance with the definition provided below.

Concomitant use of another preventive drug or use of it in less than 5-half lives of the drug.

History of another active primary headache with a periodicity considered frequent according to the International Classification of Headache disorders, that is, more than 10 days per month at the time of screening or the basal period.

Continuous or daily headache in the month prior to inclusion in the study. Pregnancy or breastfeeding. Any relevant cardiovascular conditions. Kidney diseases. Hyperkaliemia. Use of another concomitant preventive. Previous use of candesartan. Current use of another Angiotensin Conversing Enzime Inhibitor or Angiotensin-II receptor antagonist.

Alcoholism or drug use.

Concomitant treatment:

The study will not interfere in the current practice, participants will receive the candesartan in the same manner and intensity if they were not enrolled in the study.

Patients will be allowed to use their usual symptomatic treatment as usual. The number of days of symptomatic treatment and the number of use of triptans will be reflected.

The concomitant drugs with potential use as a preventive according to National Clinical Practice guidelines (gabapentin, pregabalin, tricyclic antidepressants, duloxetine, valproic acid, phenytoin, lamotrigine, topiramate, botulinum toxin, anti-CGRP antibodies, beta-blockers, lisinopril) will not be permitted.

Treatment failure shall be defined as insufficient efficacy at a sufficient dose and for an adequate duration or withdrawal due to adverse effects of a drug present in the national headache guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with episodic migraine or chronic migraine according to The International Classification of Headache Disorders, receiving Candesartan under the criteria of their physician and according to local guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Response prediction. | Weeks 20 to 24 compared with baseline period
  To determine which demographic or clinical variables present at baseline are associated with a 50% reduction in the frequency of headache days per month between weeks 20 to 24 compared with baseline in a regression analysis.

SECONDARY OUTCOMES:
Response predictors | Between weeks 20 to 24 compared with baseline period
  To determine which demographic and clinical variables present at baseline are associated with a greater reduction in the frequency of headache days per month between weeks 20 to 24 compared with baseline in a regression analysis.
Adverse events. | through study completion, an average of 24 weeks.
  To determine frequency and type of adverse effects related with candesartan through study completion, an average of 24 weeks.
Discontinuation due to adverse events. | through study completion, an average of 24 weeks.
  To evaluate percentage of patients that discontinues candesartan due to adverse events through study completion, an average of 24 weeks.
50% response rate at 24 weeks | Between weeks 20 to 24 compared with baseline period
  To evaluate percentage of patients that present a 50% response rate to candesartan in headache day reduction evaluated in the period between weeks 20 to 24 compared with baseline.
30% response rate at 24 weeks | Between weeks 20 to 24 compared with baseline period
  To evaluate percentage of patients that present a 30% response rate to candesartan in headache day reduction evaluated in the period between weeks 20 to 24 compared with baseline.
75% response rate at 24 weeks | Between weeks 20 to 24 compared with baseline period
  To evaluate percentage of patients that present a 75% response rate to candesartan in headache day reduction evaluated in the period between weeks 20 to 24 compared with baseline.
100% response rate at 24 weeks | Between weeks 20 to 24 compared with baseline period
  To evaluate percentage of patients that present a 100% response rate to candesartan in headache day reduction evaluated in the period between weeks 20 to 24 compared with baseline.
50% response rate at 12 weeks | Between weeks 8 to 12 compared with baseline period
  To evaluate percentage of patients that present a 50% response rate to candesartan in headache day reduction evaluated in the period between weeks 8 to 12 compared with baseline.
30% response rate at 12 weeks | Between weeks 8 to 12 compared with baseline period
  To evaluate percentage of patients that present a 30% response rate to candesartan in headache day reduction evaluated in the period between weeks 8 to 12 compared with baseline.
75% response rate at 12 weeks | Between weeks 8 to 12 compared with baseline period
  To evaluate percentage of patients that present a 75% response rate to candesartan in headache day reduction evaluated in the period between weeks 8 to 12 compared with baseline.
100% response rate at 12 weeks | Between weeks 8 to 12 compared with baseline period
  To evaluate percentage of patients that present a 100% response rate to candesartan in headache day reduction evaluated in the period between weeks 8 to 12 compared with baseline.
Headache days reduction at 24 weeks | Between weeks 20 to 24 compared with baseline period
  To evaluate headache days reduction in the period between weeks 20 to 24 compared with baseline.
Intense headache days reduction at 24 weeks | Between weeks 20 to 24 compared with baseline period
  To evaluate intense headache days reduction in the period between weeks 20 to 24 compared with baseline.
Acute headache medication reduction at 24 weeks | Between weeks 20 to 24 compared with baseline period
  To evaluate acute headache medication days reduction in the period between weeks 20 to 24 compared with baseline.
Headache days reduction at 12 weeks | Between weeks 8 to 12 compared with baseline period
  To evaluate headache days reduction in the period between weeks 8 to 12 compared with baseline.
Intense headache days reduction at 12 weeks | Between weeks 8 to 12 compared with baseline period
  To evaluate Intense headache days reduction in the period between weeks 8 to 12 compared with baseline.
Acute headache medication reduction at 12 weeks | Between weeks 8 to 12 compared with baseline period
  To evaluate acute headache medication days reduction in the period between weeks 8 to 12 compared with baseline.
Change in HIT-6 scale at 24 weeks | Between weeks 20 to 24 compared with baseline period
  To evaluate change in HIT-6 scale in the period between weeks 20 to 24 compared with baseline.
Change in HADS scale at 24 weeks | Between weeks 20 to 24 compared with baseline period
  To evaluate change in HADS scale in the period between weeks 20 to 24 compared with baseline.
Change in HADS scale at 12 weeks | Between weeks 8 to 12 compared with baseline period
  To evaluate change in HADS scale in the period between weeks 8 to 12 compared with baseline.
Change in heart rate at 24 weeks | Between weeks 20 to 24 compared with baseline period
  To evaluate change in heart rate (in beats per minute) in the period between weeks 20 to 24 compared with baseline.
Change in heart rate at 12 weeks | Between weeks 8 to 12 compared with baseline period
  To evaluate change in heart rate (in beats per minute) in the period between weeks 8 to 12 compared with baseline.
Change in systolic blood pressure at 24 weeks | Between weeks 20 to 24 compared with baseline period
  To evaluate change in systolic blood pressure (mmHg) in the period between weeks 20 to 24 compared with baseline.
Change in systolic blood pressure at 12 weeks | Between weeks 8 to 12 compared with baseline period
  To evaluate change in systolic blood pressure (mmHg) in the period between weeks8 to 12 compared with baseline.
Change in diastolic blood pressure at 24 weeks | Between weeks 20 to 24 compared with baseline period
  To evaluate change in diastolic blood pressure (mmHg) in the period between weeks 20 to 24 compared with baseline.
Change in diastolic blood pressure at 12 weeks | Between weeks 8 to 12 compared with baseline period
  To evaluate change in diastolic blood pressure (mmHg) in the period between weeks 8 to 12 compared with baseline.
Change in HIT-6 scale at 12 weeks | Between weeks 8 to 12 compared with baseline period
  To evaluate change in HIT-6 scale in the period between weeks 8 to 12 compared with baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario Valladolid, Valladolid, Spain

REFERENCES:
- [Background] GBD 2016 Neurology Collaborators. Global, regional, and national burden of neurological disorders, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 May;18(5):459-480. doi: 10.1016/S1474-4422(18)30499-X. Epub 2019 Mar 14. PMID 30879893
- [Background] Stovner LJ, Andree C. Prevalence of headache in Europe: a review for the Eurolight project. J Headache Pain. 2010 Aug;11(4):289-99. doi: 10.1007/s10194-010-0217-0. Epub 2010 May 16. PMID 20473702
- [Background] GBD 2017 DALYs and HALE Collaborators. Global, regional, and national disability-adjusted life-years (DALYs) for 359 diseases and injuries and healthy life expectancy (HALE) for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1859-1922. doi: 10.1016/S0140-6736(18)32335-3. PMID 30415748
- [Background] Pedraza MI, Mulero P, Ruiz M, de la Cruz C, Herrero S, Guerrero AL. Characteristics of the first 2,000 patients registered in a specialist headache clinic. Neurologia. 2015 May;30(4):208-13. doi: 10.1016/j.nrl.2013.12.010. Epub 2014 Jan 30. English, Spanish. PMID 24485650
- [Background] Evers S, Afra J, Frese A, Goadsby PJ, Linde M, May A, Sandor PS; European Federation of Neurological Societies. EFNS guideline on the drug treatment of migraine--revised report of an EFNS task force. Eur J Neurol. 2009 Sep;16(9):968-81. doi: 10.1111/j.1468-1331.2009.02748.x. PMID 19708964
- [Background] Tronvik E, Stovner LJ, Helde G, Sand T, Bovim G. Prophylactic treatment of migraine with an angiotensin II receptor blocker: a randomized controlled trial. JAMA. 2003 Jan 1;289(1):65-9. doi: 10.1001/jama.289.1.65. PMID 12503978
- [Background] Stovner LJ, Linde M, Gravdahl GB, Tronvik E, Aamodt AH, Sand T, Hagen K. A comparative study of candesartan versus propranolol for migraine prophylaxis: A randomised, triple-blind, placebo-controlled, double cross-over study. Cephalalgia. 2014 Jun;34(7):523-32. doi: 10.1177/0333102413515348. Epub 2013 Dec 11. PMID 24335848
- [Background] Garcia-Azorin D, Santos-Lasaosa S, Gago-Veiga AB, Viguera Romero J, Guerrero-Peral AL. Real world preventative drug management of migraine among Spanish neurologists. J Headache Pain. 2019 Feb 15;20(1):19. doi: 10.1186/s10194-019-0971-6. PMID 30770719
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Derived] Garcia-Azorin D, Martinez-Badillo C, Camina Muniz J, Gago-Veiga AB, Morollon Sanchez N, Gonzalez-Quintanilla V, Porta-Etessam J, Sierra-Mencia A, Gonzalez-Garcia N, Gonzalez-Osorio Y, Polanco-Fernandez M, Recio-Garcia A, Belvis Nieto R, Guerrero-Peral AL. CandeSpartan Study: Candesartan Spanish Response-prediction and Tolerability study in migraine. Cephalalgia. 2024 Apr;44(4):3331024241248833. doi: 10.1177/03331024241248833. PMID 38663908